CLINICAL TRIAL: NCT02116660
Title: Switching From Regimens Consisting of a RTV-Boosted Protease Inhibitor Plus TDF/FTC to a Combination of Raltegravir Plus Nevirapine and Lamivudine in HIV Patients With Suppressed Viremia and Impaired Renal Function (RANIA Study) (Pilot Study) Protocol MK-0518-284-03
Brief Title: Evaluation of Renal Function, Efficacy, and Safety When Switching From Tenofovir/Emtricitabine Plus a Protease Inhibitor/Ritonavir, to a Combination of Raltegravir (MK-0518) Plus Nevirapine Plus Lamivudine in HIV-1 Participants With Suppressed Viremia and Impaired Renal Function (MK-0518-284)
Acronym: RANIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to poor recruitment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0518-284; 2013-001637-40 (EudraCT Number); MK-0518-284 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Nevirapine; Lamivudine; Tenofovir; Emtricitabine; Lopinavir; Ritonavir; Atazanavir Sulfate; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raltegravir plus Nevirapine plus Lamivudine (Experimental): Raltegravir 400 mg oral twice daily for 96 weeks; plus nevirapine 200 mg oral once daily for 14 days followed by nevirapine 200 mg oral twice daily, plus lamivudine 150 mg oral twice daily for 96 weeks
  Interventions: Drug: Raltegravir (MK-0518); Drug: Nevirapine; Drug: Lamivudine
- Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine (Active Comparator): Tenofovir/emtricitabine 300/200 mg oral once daily plus 1) lopinavir/ritonavir 400/100 mg oral twice daily or 800/200 mg oral once daily, or 2) atazanavir/ritonavir 300/100 mg oral once daily, or 3) darunavir/ritonavir 800/100 mg oral once daily or 600/100 mg oral twice daily
  Interventions: Drug: Tenofovir; Drug: Emtricitabine; Drug: Lopinavir; Drug: Ritonavir; Drug: Atazanavir; Drug: Darunavir

INTERVENTIONS:
Drug: Raltegravir (MK-0518) — Raltegravir (MK-0518) 400 mg tablets
  Arms: Raltegravir plus Nevirapine plus Lamivudine
Drug: Nevirapine — Nevirapine (NVP) 200 mg tablets
  Arms: Raltegravir plus Nevirapine plus Lamivudine
Drug: Lamivudine — Lamivudine (3TC) 150 mg tablets
  Arms: Raltegravir plus Nevirapine plus Lamivudine
Drug: Tenofovir — Tenofovir disoproxil fumarate (TDF) 300 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine
Drug: Emtricitabine — Emtricitabine (FTC) 200 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine
Drug: Lopinavir — Lopinavir (LPV) 200 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine
Drug: Ritonavir — Ritonavir (r) 100 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine
Drug: Atazanavir — Atazanavir (ATV) 300 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine
Drug: Darunavir — Darunavir (DAR) 400 mg tablets
  Arms: Protease Inhibitor/Ritonavir plus tenofovir/emtricitabine

SUMMARY:
To evaluate changes in renal function, efficacy, and safety when switching from a combination of tenofovir/emtricitabine (TDF/FTC) plus a protease inhibitor/ritonavir (PI/r) to a combination of raltegravir (MK-0518) plus nevirapine plus lamivudine in human immunodeficiency virus (HIV)-1 infected participants with suppressed viremia and impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male, or non-pregnant, non-breastfeeding female
* No previous history of virological failure
* No previous exposure to non-nucleoside reverse transcriptase inhibitors or integrase inhibitors
* No previous history of intolerance to lamivudine
* At least 2 documented plasma HIV-1 RNA <50 copies/mL and no HIV-1 >50 copies/mL in the 12 months before screening
* Receiving the same protease inhibitor/ritonavir plus tenofovir/emtricitabine combination for at least the 6 months before screening
* Has no major International Antiviral Society (IAS)-USA mutations on genotype testing performed before starting antiretroviral treatment
* Sexually-active participants and their partners of child-bearing potential agree to use a medically acceptable method of contraception from 2 weeks before Day 1 and for at least 6 months after the last dose of study drug (postmenopausal women are not required to use contraception; sexually-active male participants with a female partner of child-bearing potential must provide written informed consent to information regarding any pregnancy)

Exclusion Criteria:

* Positive for hepatitis B surface antigen (HBsAg+) or anticipated need for hepatitis C virus treatment
* Liver cirrhosis
* Has a history of diabetes mellitus, defined as initiation of antidiabetic treatment or verification of diabetes in a case report form
* Has any cancer, excluding stable Kaposi Sarcoma
* Allergy or sensitivity to the investigational product or excipients
* Female participant who is nursing
* Female participant who is pregnant or intends to become pregnant
* Has an active Acquired Immunodeficiency Syndrome (AIDS)-defining event except stable Kaposi Sarcoma or HIV Wasting Syndrome
* Received any investigational drug within 30 days before screening
* Participated in any other clinical trial within 30 days before signing informed consent for the current trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Human immunodeficiency virus (HIV) infected adults with stable suppressed HIV-1 ribonucleic acid (RNA) from at least 12 months prior to the screening visit, and with a current stable anti-retroviral (ARV) regimen were enrolled in this trial.
Groups:
- Raltegravir Plus Nevirapine Plus Lamivudine: Raltegravir 400 mg orally twice daily for 96 weeks; plus nevirapine 200 mg orally once daily for 14 days followed by nevirapine 200 mg orally twice daily, plus lamivudine 150 mg orally twice daily for 96 weeks
- Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine: Tenofovir/emtricitabine 300/200 mg orally once daily plus 1) lopinavir/ritonavir 400/100 mg orally twice daily or 800/200 mg orally once daily, or 2) atazanavir/ritonavir 300/100 mg orally once daily, or 3) darunavir/ritonavir 800/100 mg orally once daily or 600/100 mg orally twice daily
Period: Overall Study
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Started | 6 | 5
Completed | 4 | 1
Not Completed | 2 | 4
Not completed — Deteriorating renal function | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Organization reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.83 (6.21) | 54.00 (5.92) | 51.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min] — Estimated Glomerular Filtration Rate (eGFR) was estimated from the Modification of Diet in Renal Disease (MDRD)-6 equation. The MDRD-6 equation = 198 × [serum creatinine(mg/dL)]^-0.858 × [age]-0.167 × [0.822 if patient is female] × [1.178 if patient is black] × [serum urea nitrogen concentration (mg/dL)]^-0.293 × [urine urea nitrogen excretion (g/d)]^0.249. Population: Data for eGFR at baseline were not determined for 1 participant in each treatment group.
  mL/min
    number analyzed (Participants) | 5 | 4 | 9
    (all) | 87.5 (7.32) | 87.7 (6.52) | 87.62 (6.54)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: Glomerular Filtration Rate (eGFR) was estimated from the Modification of Diet in Renal Disease (MDRD)-6 equation. The MDRD-6 equation = 198 × [serum creatinine(mg/dL)]^-0.858 × [age]-0.167 × [0.822 if patient is female] × [1.178 if patient is black] × [serum urea nitrogen concentration (mg/dL)]^-0.293 × [urine urea nitrogen excretion (g/d)]^0.249.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least one dose of study medications and who had both a baseline assessment, and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 5 | 4
mL/min | -1.1 (4.65) | -5.5 (11.78)

2. Secondary Outcome: Percentage of Participants With Suppressed Viremia (<50 Copies/mL HIV-1 Ribonucleic Acid [RNA]) at Week 48
Description: Plasma was to be collected at Week 48 in order to quantify HIV-1 RNA. and identify the percentage of participants with <50 copies/mL HIV-1 RNA.
Time Frame: Week 48
Population: Due to poor enrollment the study was terminated early; therefore data for secondary outcome measures were not collected, and were not analyzed.
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Suppressed Viremia (<50 Copies/mL HIV-1 RNA) at Week 96
Description: Plasma was to be collected at Week 96 in order to quantify HIV-1 RNA. and identify the percentage of participants with <50 copies/mL HIV-1 RNA.
Time Frame: Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Decline in Renal Function at Week 48
Description: Decline in renal function was to be assessed by evaluating MDRD-6, creatinine clearance and serum phosphate.
Time Frame: Week 48
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Virologic Failure (HIV-1 RNA > 50 Copies/mL)
Description: Plasma was to be collected up to Week 96 in order to quantify HIV-1 RNA, and identify the percentage of participants with >50 copies/mL HIV-1 RNA.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline of HIV-RNA Absolute Values
Description: Plasma was to be collected at baseline and Week 96 in order to determine the change from baseline in HIV-1 RNA.
Time Frame: Baseline and Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Mutations Associated With Resistance to NRTIs, NNRTIs, INI, at Virological Failure.
Description: Participants were to be identified with mutations associated with Nucleoside/ Nucleotide Reverse Transcriptase Inhibitors (NRTIs), Non-nucleoside Reverse Transcriptase Inhibitors (NNRTIs), and Integrase Inhibitor (INI). Virological failure is defined as 2 consecutive plasma HIV-1 RNA >200 copies/mL at least two weeks apart while on previous or current ARV therapy.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Absolute CD4+ T-lymphocyte Count
Description: Cluster of Differentiation 4 + (CD4+) T-lymphocyte cell counts were to be determined at baseline and Week 96, in order to determine the change from baseline.
Time Frame: Baseline and Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Altered Liver Enzymes and Lipid Profile
Description: Values of liver enzymes and lipids were to be determined from laboratory tests, in order to identify the percentage of participants classified with altered values.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With Altered Values of Tubular Kidney Injury Markers.
Description: Values of tubular kidney injury markers. were to be determined, in order to identify the percentage of participants classified with altered values.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants Having Changes From Baseline in Metabolic Bone Markers
Description: Changes from baseline in metabolic bone markers, serum Bone Specific Alkaline Phosphatase (s-BSAP) and C-telopeptides of type 1 Collagen (s-CTx), were to be determined, in order to classify the percentage of participants with changes.
Time Frame: Baseline and up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 the Last Measurement Time t (AUC0-t) for Raltegravir and Nevirapine
Description: Blood samples were to be collected in Week 12 in order to use the trapezoidal method to determine the AUC0-t of Raltegravir and Nevirapine
Time Frame: Week 12: Fasted state (0 h) and 1, 2, 3, 6 and 12 h post-dose
Population: as for outcome 2
Groups:
- Raltegravir; Nevirapine: Raltegravir 400 mg orally twice daily for 96 weeks; plus nevirapine 200 mg orally once daily for 14 days followed by nevirapine 200 mg orally twice daily, plus lamivudine 150 mg orally twice daily for 96 weeks
Arm/Group | Raltegravir | Nevirapine
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Trough Concentration (Ctrough) for Raltegravir and Nevirapine
Description: Blood samples were to be collected in Weeks 12 and 48 in order to use the trapezoidal method to determine the Ctrough, the lowest concentration reached by the drug before the next dose is administered, of Raltegravir and Nevirapine.
Time Frame: Weeks 12 and 48: at the end of dosing interval at 12 h
Population: as for outcome 2
Arm/Group | Raltegravir | Nevirapine
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Participants With Genotypic Resistance at Virologic Failure.
Description: Genotypic resistance measures the presence of particular HIV-1 mutations that give rise to drug resistance. Virological failure is defined as 2 consecutive plasma HIV-1 RNA >200 copies/mL at least two weeks apart while on previous or current ARV therapy.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Participants With Adherence to Study Therapy
Description: An Adherence Questionnaire was to be given in order to determine the percentage of participants who adhered to study therapy.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Bone Disease Risk Assessment
Description: Bone disease risk assessment was to be based on a Fracture Risk Assessment Tool (FRAX®) score in participants > 40 years old, and the change from baseline determined.
Time Frame: Baseline and week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline in the VACS Index
Description: The Veterans Aging Cohort Risk Index (VACS Index) combines various clinical biomarkers into a cumulative index weighted according to the risk of all-cause mortality.
Time Frame: Baseline and week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percentage of Participants Experiencing a Decline of Renal Function
Description: Decline in renal function was to be assessed by evaluating MDRD-6, creatinine clearance and serum phosphate.
Time Frame: Up to Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Change From Baseline in eGFR at Week 96
Description: as for outcome 1
Time Frame: Baseline and Week 96
Population: as for outcome 2
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 98
Description: All randomized participants who received at least one dose of study treatment.
Arm/Group | Raltegravir Plus Nevirapine Plus Lamivudine | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 3/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir Plus Nevirapine Plus Lamivudine (N=6) | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine (N=5)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir Plus Nevirapine Plus Lamivudine (N=6) | Protease Inhibitor/Ritonavir Plus Tenofovir/Emtricitabine (N=5)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02116660/Prot_SAP_000.pdf